CLINICAL TRIAL: NCT06410963
Title: ReActivate: Physiotherapist Led Intervention for Adolescents With Pain and Psychological Distress. A Sequential Replicated and Randomized Single Case Experimental Design (SCED).
Brief Title: ReActivate: Physiotherapist Led Intervention for Adolescents With Pain and Psychological Distress.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Reactivate
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain; Emotional Distress
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This study employs a sequential single-case experimental AB design with randomized waiting period lengths (7, 14 or 21 days). Included in the design is also standardized pre-post and 6-month follow up measurement allowing for single group analysis of change. In addition, we collect qualitative data from participating adolescents.
Who Masked: Outcomes Assessor
Masking Description: Data is collected using a secure digital platform. Outcome assessors will be blinded to baseline length allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No treatment waiting period (No Intervention): Participants are randomized to a 7, 14 or 21 day waiting period. Daily measurements are collected throughout this period.
- Reactivate (Experimental): Reactivate treatment. Daily measurements are collected throughout treatment.
  Interventions: Behavioral: Reactivate

INTERVENTIONS:
Behavioral: Reactivate — The study period is 84 days (12 weeks). Depending on the length of the baseline period (randomly assigned to be 7, 14 or 21 days), the treatment period varies between 63-77 days and contains 6-11 sessions. The intervention consists of 2-4 educational sessions in pain mechanisms and fear avoidance and 4-9 sessions of individually tailored intervention with graded exposure and reactivation to avoided physical activities. Intervention will take place from one time per week to one time every two weeks, 30-60 minutes per session. Number of treatment sessions will depend on when the individual participants' goals are considered reached. If necessary, given the participants consent, their legal guardians will be invited to attend the sessions.
  Arms: Reactivate

SUMMARY:
Recurrent or persistent pain and psychological distress are alarmingly common problems among adolescents, in Sweden as well as globally. They often co-occur and have been shown to be predictors of sustained problems in adulthood. Adequate treatment early on in the development of problems has been shown important in order to decrease the risk of sustained problems in adulthood but available treatments have only modest effects. There is thus a need for treatment development, not in the least for (secondary) preventative purposes. The aim of this project is therefore to develop an evidence based and cost-effective secondary preventative intervention. Specifically, this project aims to develop and test a physiotherapist led treatment for adolescents with recurrent or persistent pain and psychological distress based upon graded exposure to physical activity and reactivation.

DETAILED DESCRIPTION:
See description of arms and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-19
* Psychological distress, such as anxiety, depressive symptoms or stress, ≥2 on a numeric rating scale 0-6 (0=not at all, 6=to a great extent)
* Persistent (consistently or weekly recurrent) musculoskeletal pain problems for ≥3 months, with pain intensity ≥2 on a numeric rating scale 0-6 (0=not at all, 6=to a great extent)
* Presence of avoidance behaviour and/or or worry about symptoms/problems, ≥1 on a numeric rating scale 0-6 (0=not at all, 6=to a great extent); > 50 on at least one activity of the PHODA.
* Swedish speaking and able to fill out questionnaires

Exclusion Criteria:

* Serious/malignant disease
* Participation in other rehabilitation program
* Severe mental health problems
* Substance abuse
* Severe learning disabilities

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Activity engagement change | repeated daily through phase A (randomly assigned to be 7, 14 or 21 days) and treatment phase B (9-11 weeks). Total time frame of assessment is 12 weeks (84 days). 7 days assessment 6 months after terminated intervention
  Change in self-rated activity engagement. Numerical Rating Scale, range 0-6 (1 question: lower values, worse outcome, 1 question: Lower values, better outcome )
Symptom distress change | repeated daily through phase A (randomly assigned to be 7, 14 or 21 days) and treatment phase B (9-11 weeks). Total time frame of assessment is 12 weeks (84 days). 7 days assessment 6 months after terminated intervention.
  Change in self-rated distress about symptoms. Numerical Rating Scale, range 0-6 (3 questions, higher values, worse outcome)

SECONDARY OUTCOMES:
Functional Disability Inventory (FDI) change | baseline, after treatment phase B (12 weeks), 6 months after terminated intervention
  Change in functional disability. Descriptive Rating Scale, range 0-64 (higher values, worse outcome)
Center of Epidemiological Studies Depression Scales for Children (CES-DC) change | baseline, after treatment phase B (12 weeks), 6 months after terminated intervention
  Change in depressive symptoms. Descriptive Rating Scale, range 0-60 (higher values, worse outcome)
The Pediatric Quality of Life Acute version (PedsQL) PedsQL™ | baseline, after treatment phase B (12 weeks), 6 months after terminated intervention
  Change in quality of life. Descriptive Rating Scale, range 0-92 (higher values, worse outcome)
Change in psychological distress | repeated daily through phase A (randomly assigned to be 7, 14 or 21 days) and treatment phase B (9-11 weeks). Total time frame of assessment is 12 weeks (84days). 7 days assessment 6 months after terminated assessment.
  Change in self-related symptoms of psychological distress. Numerical Rating Scale, range 0-6 (3 questions, higher values, worse outcome)
Pain change | repeated daily through phase A (randomly assigned to be 7, 14 or 21 days) and treatment phase B (9-11 weeks). Total time frame of assessment is 12 weeks (84days). 7 days assessment 6 months after terminated assessment.
  Change in self-related pain symptoms. Numerical Rating Scale range 0-6 (higher values, worse outcome)
Fear of Pain Questionnaire Children Short-form (FOPQ-C SF) change | baseline, after treatment phase B (12 weeks), 6 months after terminated intervention
  Change in fear of pain. Descriptiv Rating Scale, range 0-40 (higher values worse outcome)
The Photograph Series of Daily Activities for youth (PHODA) change - short | First session after baseline (randomly assigned to be 7, 14 or 21 days), after treatment phase B (12 weeks)
  Change in percieved harmfulness. Photographs with 50 activities, rated on a Subjective Self-rating Scale, range 0-100mm/item (higher values, worse outcome)

OTHER OUTCOMES:
Treatment Inventory of Costs in Patients with psychiatric disorders (Tic-P), medical resources | baseline, 12 weeks, 6 months after terminated intervention
  Change in use of medical resources. Dichotomous scale completed by open ended answers if answer is yes.
Treatment Inventory of Costs in Patients with psychiatric disorders (Tic-P), school absence | baseline, 12 weeks, 6 months after terminated intervention
  Change in school abcense. Dichotomous scale completed by open ended answers if answer is yes. One question is completed by one question with Numerical Rating Scale 1-10 (higher values, worse outcome) if answer is yes.
Accelerometer | 7 days of the first week of baseline (randomly assigned to be 7, 14 or 21 days). 7 days assessment 6 months after terminated assessment.
  Change in physical activity, digital device counting steps

CONTACTS AND LOCATIONS:
Overall Officials: Katja Boersma, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Region Örebro county, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No